CLINICAL TRIAL: NCT04595994
Title: Phase I/II Randomized Clinical Trial of Selinexor Plus Gemcitabine in Selected Advanced Soft-tissue Sarcoma and Osteosarcoma
Brief Title: Selinexor Plus Gemcitabine in Selected Advanced Soft-tissue Sarcoma and Osteosarcoma
Acronym: SeliSarc
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-67; 2019-000652-33 (EudraCT Number)
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — selinexor; Gemcitabine

STUDY DESIGN:
Intervention Model Description: unique arms for each possible dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor + Gemcitabine (Experimental): Dose escalation levels (Phase I):
  All included patients will take both drugs:
  Selinexor weekly (given on days 1,8 and 15 of each cycle) will be dispensed at different dose levels: dose level 1:60 mg, dose level 2: 60 mg, dose level 3: 60 mg, and dose level 4: 80 mg).
  Gemcitabine weekly (given on days 1, 8 of each cycle) will be administered at different dose levels: (dose level 1:1000 mg/m2 (30 min), dose level 2:1000 mg/m2 (10 mg/m2/min), dose level 3:1200 mg/m2 (10 mg/m2/min) and dose level 4: 1200 mg/m2 (10 mg/m2/min)).
  Selinexor: tablet (20 mg tablets) Oral use.
  Gemcitabine: Concentrate for solution for infusion. Intravenous use.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — For both interventional ( Selinexor and Gencitabine) Dose-limiting toxicity (DLT) will be applied only to either of the following toxicities occurring during the first treatment cycle (days 1-21).
  Other Names: Gemcitabine

SUMMARY:
Phase I-II, randomized, open-label, multicenter, international clinical trial Patients with advanced soft-tissue sarcoma (undifferentiated pleomorphic sarcoma, leiomyosarcoma, alveolar soft-part sarcoma) and osteosarcoma will receive selinexor in combination with gemcitabine.

DETAILED DESCRIPTION:
Phase I-II, randomized, open-label, multicenter, international clinical trial Patients with advanced soft-tissue sarcoma (undifferentiated pleomorphic sarcoma, leiomyosarcoma, alveolar soft-part sarcoma) and osteosarcoma will receive selinexor in combination with gemcitabine.

In the Phase I part safety and toxicity of the combination will be assessed using a 3+3 design. The recommended dose for the Phase II will be determined.

In the Phase II part there will be 4 different cohorts:

Cohort 1: Undifferentiated pleomorphic sarcoma (UPS) Cohort 2: Leiomyosarcoma (LMS) Cohort 3: Alveolar soft-part sarcoma (ASPS) Cohort 4: Osteosarcoma Patients will be randomized for phase II part only (except in cohort 3) in an open-label way to receive selinexor in combination with gemcitabine versus gemcitabine alone

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of any study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. imaging tests), obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 18-80 years
3. Histologic diagnosis of soft tissue sarcoma (undifferentiated pleomorphic sarcoma, leiomyosarcoma, alveolar soft part sarcoma) or osteosarcoma confirmed by central pathology review prior to enrolment with an archive tumor sample. A fresh paraffin embedded tumor tissue block must be provided for all subjects for biomarker analysis before and (when feasible) after treatment with investigational products.
4. Metastatic/advanced disease in progression in the last 6 months.
5. Patients have previously received at least one previous line of systemic therapy
6. Measurable disease according to RECIST 1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. Adequate hepatic, renal, cardiac, and hematologic function.
9. Laboratory tests as follows:

   * Absolute neutrophil count ≥ 1,500/mm³
   * Platelet count ≥ 100,000/mm³
   * Bilirubin ≤ 1.5 mg/dL
   * AST and ALT ≤ 2.5 times upper limit of normal
   * Creatinine ≤ 1.5 mg/dL
10. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan.
11. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to enrollment and agree to use birth control measures during study treatment and for 3 months after its completion. Patients must not be pregnant or nursing at study entry. Women/men of reproductive potential must have agreed to use an effective contraceptive method.

Exclusion Criteria:

1. Three or more previous lines of chemotherapy
2. Prior selinexor or another XPO1 inhibitor treatment.
3. Administration of a previous gemcitabine-containing treatment.
4. Any concurrent medical condition or disease (e.g. uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
5. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
6. Pregnant or breastfeeding females.
7. Body surface area (BSA) <1.4 m2 at baseline, calculated by the Du Bois(31) or osteller(32) method.
8. Life expectancy of less than 3 months.
9. Major surgery within 4 weeks prior to C1D1.
10. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or dysfunction that could interfere with absorption of study treatment.
11. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the NCCN CPGO for antiemesis and anorexia/cachexia (palliative care).
12. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
13. Presence of brain or central nervous system metastases, unless they are controlled (patients with treated and stable metastasis are eligible).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 6 months
  To determine the maximum tolerated dose (MTD) or the recommended dose for phase II of Selinexor plus gemcitabine.

SECONDARY OUTCOMES:
Safety profile according to CTCAE 5.0. | 6 months
  Safety profile of the experimental treatment, through assessment of adverse event type, incidence, severity, time of appearance, related causes, as well as physical explorations and laboratory tests.
Objective response rate (ORR). | 6 months
  Objective Response Rate (ORR): ORR is defined as the number of subjects with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) divided by the number of response evaluable subjects (according to RECIST 1.1 criteria).
Evaluate efficacy according to Choi response | 6 months
  Efficacy measured through tumor response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression.
Patients's quality of life (QoL) | 6 months
  Quality of life will be measured with European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire 30
Pharmacokinetic values in blood analysis | 6 months
  Impact of pharmacokinetics. interactions between selinexor in gemcitabine

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín Broto, MD, Study Director — Hospital Fundación Jiménez Díaz
Locations (6):
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - HU Vall d'Hebron, Barcelona
  - H. Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kashyap T, Argueta C, Unger T, Klebanov B, Debler S, Senapedis W, Crochiere ML, Lee MS, Kauffman M, Shacham S, Landesman Y. Selinexor reduces the expression of DNA damage repair proteins and sensitizes cancer cells to DNA damaging agents. Oncotarget. 2018 Jul 20;9(56):30773-30786. doi: 10.18632/oncotarget.25637. eCollection 2018 Jul 20. PMID 30112106
- [Background] Park KS, Han BG, Lee KH, Kim DS, Kim JM, Jeon H, Kim HS, Suh SW, Lee EH, Kim SY, Lee BI. Depletion of nucleophosmin via transglutaminase 2 cross-linking increases drug resistance in cancer cells. Cancer Lett. 2009 Feb 18;274(2):201-7. doi: 10.1016/j.canlet.2008.09.007. Epub 2008 Oct 11. PMID 18851895
- [Background] Hill R, Rabb M, Madureira PA, Clements D, Gujar SA, Waisman DM, Giacomantonio CA, Lee PW. Gemcitabine-mediated tumour regression and p53-dependent gene expression: implications for colon and pancreatic cancer therapy. Cell Death Dis. 2013 Sep 5;4(9):e791. doi: 10.1038/cddis.2013.307. PMID 24008735
- [Derived] Martin-Broto J, Casado A, Marquina G, Redondo A, Martinez-Trufero J, Valverde C, Gutierrez A, Bernabeu D, Ortega L, Merino J, Ramos R, Ledesma P, Mondaza-Hernandez JL, Moura DS, Hindi N. Gemcitabine plus selinexor in selective advanced sarcomas: a phase I of the Spanish group for research on sarcoma study. Nat Commun. 2026 Jan 20. doi: 10.1038/s41467-026-68729-1. Online ahead of print. PMID 41559089